CLINICAL TRIAL: NCT05837624
Title: Estetrol/Drospirenone to Reduce the Average Size of Endometriomas
Acronym: ERASE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Andrew Zakhari (Other)
Responsible Party: Sponsor-Investigator, Andrew Zakhari, Dr. Andrew Zakhari, MD, FRCSC, MGSC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-9147
Record Dates: First submitted 2023-04-12; First posted 2023-05-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Endometrioma; Endometrioma
Keywords: Estetrol/drospirenone; Nextstellis; Endometriosis; volume reduction; ultrasound; Estetrol-drospirenone
MeSH Terms: conditions — Endometriosis | interventions — drospirenone and estetrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women with an ovarian endometrioma who will take drospirenone / estetrol (Experimental): Women 18 years of age or older with endometriosis who have at least one ovarian endometrioma, of at least 3 cm in diameter, who will take oral Drospirenone / Estetrol treatment for 6 months
  Interventions: Drug: Estetrol/Drospirenone

INTERVENTIONS:
Drug: Estetrol/Drospirenone — 6-month course of oral estetrol/drospirenone (15 mg estetrol monohydrate / 3 mg drospirenone) once daily for the study duration

SUMMARY:
Endometriosis, a chronic gynecological disorder associated with pain and infertility, is a common condition affecting approximately one in ten women. Up to 50% of patients with endometriosis have ovarian endometriomas (or "chocolate cysts"). These cysts directly impact fertility and ovarian reserve (ie. ability to have children) and can cause additional symptoms in women such as added pain, discomfort, and surgical emergencies (cyst rupture, or more rarely twisting). While endometriomas tend to require surgical excision as a solution, medical management with a variety of medications has been shown to be effective in reducing their size.

Medical management (ie. medications and treatments that don't involve surgery) to reduce cyst size can help relieve symptoms either as a long term solution, before fertility treatments, or temporarily until surgery can be offered. Because the COVID-19 pandemic caused significantly reduced access to surgery and resources, medical management has become important for relief of the overburdened healthcare network.

The purpose of this study is to see how effective Estetrol/drospirenone, a combined oral contraceptive (COC), is in the reduction of ovarian endometriomas after a 3- and 6-month period of treatment.

This single arm interventional study will recruit women 18 years or older with an ovarian endometrioma of at least 3cm, who are seeking a hormonal treatment for their endometrioma(s). Consenting participants of the study will take Estetrol/drospirenone once daily, orally, for a 6 month duration. An ultrasound assessment of ovarian endometrioma(s) will be performed before starting the drug (0 months), and will be repeated at 3-months and 6-months time. At each of these hospital visits (0, 3 & 6 months), participants will have their weight and blood pressure measured, and they will complete questionnaires regarding their endometriosis symptoms, incidence of amenorrhea, compliance and incidence of any adverse effects.

DETAILED DESCRIPTION:
Ovarian endometriomas (or "chocolate cysts") are present in up to 50% of patients with endometriosis - a chronic gynecological disorder associated with pain and infertility. These cysts directly impact fertility and ovarian reserve and can cause additional symptoms in women such as added pain, discomfort, and surgical emergencies (cyst rupture, or more rarely torsion).

While endometriomas tend to require surgical excision for definitive resolution, medical management with a variety of agents has been shown to be effective in reducing their size; these agents include combined oral contraceptives (COC), aromatase inhibitors, progestins, androgens, cabergoline, and gonadotropin-releasing hormone agonists (GnRH-a). Medical management to reduce their size can help alleviate symptoms indefinitely without damaging ovarian reserve prior to fertility treatments, or to temporize until surgical management can be offered. Medical management has become particularly important in light of the COVID-19 pandemic, with significantly reduced access to surgery, and resource allocation to alleviate an overburdened healthcare network.

Estetrol/drospirenone (Nextstellis™) is a prescription-only COC available in Canada containing two hormones: a progestin (drospirenone - well known as both a standalone contraceptive and in other combined formulations), and an estrogen (estetrol - newly introduced with this product). While ethinyl estradiol (EE) is the most common estrogen currently used in COC, estetrol (E4) has proven safety and tolerability, and emerging evidence points towards a lower risk of thrombosis than traditional EE used in other COC. Studies have documented efficacy and safety for the combination estetrol/drospirenone, with a favourable bleeding profile, and very low rates of adverse reactions. While there exists already encouraging data on drospirenone and drospirenone containing products on alleviating symptoms of endometriosis and reducing the size of endometriomas, there are no studies to date evaluating this novel combination of estetrol/drospirenone in managing ovarian endometriomas.

The primary objective of this study is to determine the effectiveness of Estetrol/drospirenone, a combined oral contraceptive (COC), in the reduction of ovarian endometriomas after a 3- and 6-month period of treatment.

This is a single-center, open label, single arm interventional study that will be performed at the McGill University Health Centre (MUHC) Royal Victoria Hospital (RVH). Women 18 years of age or older with at least one ovarian endometrioma, of at least 3cm, who are seeking a hormonal treatment for their endometrioma(s), will be recruited. The study will aim to recruit 21 women.

Consenting participants will be given a 6-month course of oral estetrol/drospirenone (15 mg estetrol monohydrate / 3 mg drospirenone) once daily for the study duration. An ultrasound assessment of ovarian endometrioma(s) will be performed prior to drug initiation (baseline), and will be repeated at 3-months and 6-months time. All ultrasounds will be performed by the same ultrasonographer using a standardized technique and 3-D volumetric assessment. At each of these hospital visits, participants will have their weight and blood pressure measured and they will complete questionnaires regarding their endometriosis symptoms with a research coordinator. Safety, tolerability, and the incidence of adverse effects will also be monitored at the same time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Equal to or greater than 18 years old
* Has at least one ovarian endometrioma, of at least 3 cm
* Seeking a hormonal treatment for their endometrioma(s)

Exclusion criteria:

* Any allergy or contraindication to the study drug
* Inability to provide informed consent
* Any hormone use, from the following list, within last 3 months (excluding hormones used for ovarian stimulation for fertility treatments): Estrogen (agonist or antagonist), Progestogen (agonist or antagonist), Androgen (agonist or antagonist), GnRH (agonist or antagonist), Cabergoline

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in ovarian endometrioma volume at 6-months (from baseline) | pre-study, 6-months of treatment
  Endometrioma volume will be assessed by the same ultrasonographer (Dr. DB Nguyen) at each hospital visit, using a standardized technique, with 3-dimensional volumetric assessment.

SECONDARY OUTCOMES:
Change in endometrioma volume at 3-months (from baseline) | pre-study, 3-months of treatment
  Endometrioma volume will be assessed by the same ultrasonographer (Dr. DB Nguyen) at each hospital visit, using a standardized technique, with 3-dimensional volumetric assessment.
change in endometrioma maximal diameter at 6-months (from baseline) | pre-study, 6-months of treatment
  Endometrioma maximal diameter will be assessed by the same ultrasonographer (Dr. DB Nguyen) at each hospital visit, using a standardized technique, with 3-dimensional volumetric assessment.
change in endometrioma maximal diameter at 3-months (from baseline) | pre-study, 3-months of treatment
  Endometrioma maximal diameter will be assessed by the same ultrasonographer (Dr. DB Nguyen) at each hospital visit, using a standardized technique, with 3-dimensional volumetric assessment.
Incidence of amenorrhea | pre-study, 3-months of treatment, 6-months of treatment
  Incidence of amenorrhea will be evaluated by having the participant complete a questionnaire at each hospital visit.
  * If they have gotten their period in the last 3 months: measured by (yes/no)
  * The frequency of spotting in the last month: measured by a 4-point likert scale (Never/Rarely/Occasionally/Often)
Change in patient reported endometriosis symptoms | pre-study, 3-months of treatment, 6-months of treatment
  Change of endometriosis symptoms will be evaluated by monitoring the changes in participants's responses to the modified Biberoglu & Behrman (B&B) scale questionnaire. This is a validated scale that evaluates endometriosis pain by patient's self-assessment of three pain symptoms (dysmenorrhea, dyspareunia, and chronic pelvic pain) on a 4-point likert scale (none=0/mild=1/moderate=2/severe=3).
  Minimum value: 0 --> best outcome Maximum value: 9 --> worst outcome
Change in weight | pre-study, 3-months of treatment, 6-months of treatment
  Weight will be measured by a research coordinator or nurse at each hospital visit.
Change in blood pressure | pre-study, 3-months of treatment, 6-months of treatment
  Blood pressure will be measured by a research coordinator or nurse at each hospital visit.
Incidence of adverse effects (safety, tolerability) | 3-months of treatment, 6-months of treatment
  Incidence of adverse effects (yes/no) including: nausea/vomiting, edema, breast tenderness, headache, cramps/bloating, mood swings (specified), as well as any unexpected adverse effects will be evaluated by having the participant complete a questionnaire at each hospital visit after starting estetrol/drospirenone.
Compliance | 3-months of treatment, 6-months of treatment
  Drug compliance will be evaluated by having the participant complete a questionnaire at each hospital visit after starting estetrol/drospirenone.
  * If they have been taking the prescribed dosage of 1 oral tablet of estetrol/drospirenone a day (yes/no)
  * If they have been taking the prescribed dosage at the same time every day (yes/no)
  * How often they miss a pill, on a 4-point likert scale (Never/Rarely/Occasionally/Often)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zakhari, M.D., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liao C, Pal L. Novel Pharmacotherapies for Menopausal Symptoms. Obstet Gynecol. 2025 Oct 1;146(4):473-486. doi: 10.1097/AOG.0000000000006025. Epub 2025 Aug 7. PMID 40773756